CLINICAL TRIAL: NCT02506114
Title: An Open Label, Randomized Phase 2 Trial of Prostvac and Ipilimumab as Monotherapy or in Combination for Men With Localized Prostate Cancer Undergoing Radical Prostatectomy
Brief Title: Neoadjuvant PROSTVAC-VF With or Without Ipilimumab for Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Lawrence Fong (Other)
Collaborators: Bavarian Nordic (Industry)
Responsible Party: Sponsor-Investigator, Lawrence Fong, Professor, Department of Medicine (Hematology/Oncology), University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14559; NCI-2017-01679 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Prostatic Neoplasms
Keywords: prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: PROSTVAC-V/F (Experimental): PROSTVAC-V: 2 x 10^8pfu; subcutaneous; Day 1. PROSTVAC-F: 1 x 10^9pfu; subcutaneous; Days 15, and 36.
  Interventions: Biological: PROSTVAC V/F
- Arm B: Ipilimumab Monotherapy (Experimental): Ipilimumab: 3 mg/kg; intravenously; Days 1 and 21.
  Interventions: Drug: Ipilimumab
- Arm C: Combined PROSTVAC-V/F + Ipilimumab (Experimental): PROSTVAC-V: 2 x 10^8pfu; subcutaneous; Day 1. PROSTVAC-F: 1 x 10^9pfu; subcutaneous; Days 15, and 36. Ipilimumab: 3 mg/kg; intravenously; Days 15 and 36.
  Interventions: Biological: PROSTVAC V/F; Drug: Ipilimumab

INTERVENTIONS:
Biological: PROSTVAC V/F — PROSTVAC-V/F is a prostate-specific antigen(PSA)-based immunization strategy. It is intended to generate immune responses to prostate specific antigens and prostate cancer cells. It uses poxviral vectors to introduce modified PSA to the patient in an immunogenic manner to break self-tolerance, and thereby induce immune responses directed against prostate cancer cells.
  Arms: Arm A: PROSTVAC-V/F; Arm C: Combined PROSTVAC-V/F + Ipilimumab
Drug: Ipilimumab
  Arms: Arm B: Ipilimumab Monotherapy; Arm C: Combined PROSTVAC-V/F + Ipilimumab

SUMMARY:
This is a multicentered, open label, randomized phase II trial of PROSTVAC or ipilimumab or the combination of PROSTVAC and ipilimumab as neoadjuvant therapy in patients with localized prostate cancer. Eligible patients will be randomized to PROSTVAC monotherapy (Arm A), ipilimumab monotherapy (Arm B), or combination therapy with both PROSTVAC and ipilimumab (Arm C), prior to RP. In arms A and C, PROSTVAC-V will be administered subcutaneously as the primary vaccine on Day 1, which will be followed 2 weeks later with a series of 2 PROSTVAC-F subcutaneous administrations, given 3 weeks apart. In arms B and C, ipilimumab will be administered twice, at a dose of 3mg/kg, 3 weeks apart. In the combination arm, ipilimumab administration will coincide with the PROSTVAC-F administration. In arm B, ipilimumab will begin on Day 1. In all three arms, radical prostatectomy (RP) will occur 21 days, or three weeks, following final treatment administration of PROSTVAC or ipilimumab. No further therapy will be administered on study following RP.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be eligible for participation in this study, all of the following criteria must be satisfied:

1. Patients must have histologically confirmed adenocarcinoma of the prostate without previous therapy for prostate cancer (PC).

   * Treatment-naïve AND
   * Undergoing radical prostatectomy (RP) as initial, locally definitive therapy for PC and
   * Eligible for RP in a 3 month timeframe AND
   * Consentable for RP
2. Subject's archival prostate biopsy specimen is available, and subject consents to provide tissue for study endpoint analysis. The prostate biopsy slides or blocks must be available prior to starting any study treatment.
3. Age ≥ 18 years
4. Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Subject has adequate organ function, defined as:

   * White blood cell (WBC) count ≥ 3,000/microliter (mcL)
   * Absolute neutrophil count (ANC) ≥ 1,500/mcL
   * Platelet count ≥ 100,000/mcL
   * Hemoglobin (Hgb) ≥ 10.0 g/dL
   * Creatinine ≤ 1.5x institutional upper limit of normal (ULN)
   * Total bilirubin ≤ 1.5 x institutional ULN
   * Alanine aminotransferase (ALT) ≤ 1.5 x institutional ULN
   * Aspartate aminotransferase (AST) ≤ 1.5 x institutional ULN
   * Prothrombin time (PT) /International Normalized Ratio (INR), partial thromboplastin time (PTT) within institutional ULN
6. No known history of human immunodeficiency virus (HIV) 1 and 2, human T-cell lymphotropic virus (HTLV)-I/II, and Hepatitis B and C.
7. Ability to understand a written informed consent document, and the willingness to sign it.
8. Because of the unknown potential risk to a gamete and/or developing embryo from these investigational therapies, subjects must agree to use adequate contraception (i.e. barrier method) for the duration of study participation, and for three months after discontinuing therapy.

Exclusion Criteria:

A subject will not be eligible for participation in this study if any of the following criteria apply.

1. Subject's biopsy specimen reveals neuroendocrine or small cell features.
2. Subject has any evidence of metastatic disease (pre-operative staging will be undertaken per urologic standard of care) as deemed by the Investigator.
3. Subject has prior use of any hormones, including luteinizing hormone-releasing hormone (LHRH) agonists, ketoconazole, antiandrogens (such as bicalutamide, flutamide, or nilutamide), or 5-α-reductase inhibitors.
4. Subject has prior use of any anti-cancer treatment or product, such as PC-SPES (or any other PC-x product: PC-HOPE, PC-CARE, PC-PLUS, etc).
5. Subject has received prior radiation therapy or chemotherapy for prostate cancer.
6. Chronic administration (defined as daily or every other day for continuous use >14 days) of systemic corticosteroids within 28 days of the first planned dose off PROSTVAC-V/F. Use of inhaled steroids, nasal sprays, and topical creams for small body areas are allowed.
7. Active atopic dermatitis or skin condition that disrupts the epidermis
8. Inflammatory eye disease requiring steroid treatment
9. History of prior solid organ or bone marrow transplant
10. Previous history of hypersensitivity to eggs or allergy or untoward reaction to prior vaccinia (smallpox) vaccination.
11. Splenectomy
12. Subject, or subject's close household contacts (defined as those who share housing or have close physical contact) have any of the following conditions during the screening and/or treatment periods:

    * active or a history of atopic dermatitis, eczema or other eczematoid skin disorders that disrupt the epidermis
    * other acute, chronic or exfoliative skin conditions (e.g., burns, impetigo, varicella zoster, severe acne or other open rashes or wounds) until condition resolves
    * pregnant or nursing
    * immunodeficient or immunosuppressed (by disease or therapy), including HIV infection
13. Subject's close household contacts include children less than the age of three
14. History of, or active autoimmune disease (e.g., autoimmune neutropenia, thrombocytopenia, or hemolytic anemia, systemic lupus erythematosis, Sjogren´s syndrome, scleroderma, myasthenia gravis, Goodpasture´s syndrome, Addison´s disease, Hashimotos´s thyroiditis, or Graves disease) as determined by the treating medical oncologist.

    * Persons with vitiligo are not excluded.
    * Diabetics are not excluded if the condition is well controlled:

      1. Hemoglobin A1C < 7.0, and
      2. No evidence of end-organ damage due to diabetes, such as diabetic retinopathy, nephropathy, or neuropathy
      3. Persons with type 2 diabetes are not excluded since this is not an autoimmune disease, and do not need to meet these criteria.
    * Persons with hypothyroidism are not excluded if condition is well controlled, and condition is due to a non-autoimmune etiology.
15. Subject has received treatment with any investigational immunotherapy within 2 years prior to study screening or has received treatment with any other investigational product within 28 days prior to study screening.
16. Subject has participated in any previous study involving PROSTVAC-V/F, Sipuleucel-T or ipilimumab, regardless of whether the subject received PROSTVAC-V/F, Sipuleucel-T or ipilimumab.
17. Subject has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to PROSTVAC-V/F or ipilimumab.
18. Subject has a history of stage III or greater cancer, excluding prostate cancer. Subjects with a history of basal or squamous cell skin cancers are allowed, provided that the subject was adequately treated and is disease-free at the time of study screening. Subjects with a history of stage I or II cancer must have been adequately treated and been disease-free for ≥ 3 years prior to study screening.
19. Subject has any uncontrolled, concurrent illness including, but not limited to the following: ongoing or active infection (bacterial, viral, or fungal), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, stroke or myocardial infarction within 6 months, or psychiatric illness that would limit compliance with study requirements.
20. Subject requires any medical intervention(s) or has any other condition(s) that, in the Investigator's opinion, will 1) make the administration of PROSTVAC or ipilimumab hazardous, 2) obscure the interpretation of adverse events (AEs), 3) compromise adherence with study requirements, or 4) otherwise compromise the study's objectives.
21. Subject has high-risk features (e.g., based on Gleason score, PSA, clinical stage, % positive biopsies), and the treating physician feels the subject should undergo radical prostatectomy sooner than planned within the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Ipilimumab Montherapy: Ipilimumab: 3 mg/kg; intravenously; Days 1 and 21.
Period: Overall Study
Arm/Group | Arm A: PROSTVAC-V/F | Arm B: Ipilimumab Montherapy | Arm C: Combined PROSTVAC-V/F + Ipilimumab
Started | 5 | 4 | 6
Completed | 5 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: PROSTVAC-V/F | Arm B: Ipilimumab Monotherapy | Arm C: Combined PROSTVAC-V/F + Ipilimumab | Total
Number analyzed (Participants) | 5 | 4 | 6 | 15
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 1 | 0 | 2 | 3
  60-69 years old | 1 | 2 | 3 | 6
  70-79 years old | 3 | 2 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 5 | 4 | 6 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 4 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 3 | 4 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 6 | 15
Total Gleason Score [Count of Participants; unit: Participants] — Gleason Scores are derived from a pathology grade assigned to cancer cells on a scale of 1 to 5. Grade 1 cells resemble normal prostate tissue and Grade 5 cells are considered "high-grade" and have mutated to the extent that they barely resemble normal cells. A pathologist will assign one Gleason grade to the most predominant pattern and a second Gleason grade to the second most predominant pattern. The two grades are added together to determine the Gleason score. Theoretically scores range from 2-10, with a score of 6=low grade, 7= intermediate grade, and 8-10 = high grade.
  Participants
    Gleason Score = 6 | 0 | 0 | 1 | 1
    Gleason Score = 7 | 3 | 1 | 4 | 8
    Gleason Score = 8 | 0 | 0 | 0 | 0
    Gleason Score = 9 | 2 | 3 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Positive CD3+ T Cell Immune Response
Description: The proportion of participants who demonstrated a positive response following neoadjuvant therapy as measured by change from baseline in CD3+ T cell infiltration within prostate tumor tissue by immunohistochemistry (IHC) assessment following treatment will be reported. The change in the number of CD3+ T cell infiltration within prostate tissue between the biopsy and radical prostatectomy (RP) specimen will be quantified using immunohistochemistry (IHC),with a positive result if there is >=2 fold increase in the number of CD3+T cell infiltration.
Time Frame: Up to 2 years
Population: Few participants had evaluable labs for this outcome.
Measure: Number; unit: proportion of participants
Arm/Group | Arm A: PROSTVAC-V/F | Arm B: Ipilimumab Monotherapy | Arm C: Combined PROSTVAC-V/F + Ipilimumab
Number analyzed (Participants) | 2 | 3 | 3
proportion of participants | 0 | 0.33 | 0

2. Secondary Outcome: Proportion of Participants With Any Positive Change in Immunologic Infiltration (CD3)
Description: The proportion of participants who demonstrated any change in the number of infiltrating T cells/μm2 of CD3 within the prostatic tumor tissue from the diagnostic core biopsy specimens to the post treatment prostatectomy tissue specimens will be assessed, based upon IHC analysis following neoadjuvant PROSTVAC, ipilimumab, or the combination of the two treatments.
Time Frame: Up to 2 years
Population: Few participants had evaluable labs for this outcome.
Measure: Number; unit: proportion of participants
Arm/Group | Arm A: PROSTVAC-V/F | Arm B: Ipilimumab Monotherapy | Arm C: Combined PROSTVAC-V/F + Ipilimumab
Number analyzed (Participants) | 2 | 3 | 3
proportion of participants | 0 | 0.667 | 0

3. Secondary Outcome: Proportion of Participants With Any Positive Change in Circulating Effector T Cells
Description: The proportion of participants who demonstrated any change in the number of circulating effector T cells/μm2 within the prostatic tumor tissue from the diagnostic core biopsy specimens to the post treatment prostatectomy tissue specimens will be assessed, based upon IHC analysis following neoadjuvant PROSTVAC, ipilimumab, or the combination by flow cytometry assessment of peripheral blood mononuclear cells
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Arm A: PROSTVAC-V/F | Arm B: Ipilimumab Monotherapy | Arm C: Combined PROSTVAC-V/F + Ipilimumab
Number analyzed (Participants) | 5 | 4 | 6
proportion of participants | 0.8 | 1.0 | 0.8333

4. Secondary Outcome: Proportion of Participants With a Positive Change in Regulatory T Cells
Description: The proportion of participants who demonstrated a change in the number of Regulatory T Cells/μm2 within the prostatic tumor tissue from the diagnostic core biopsy specimens to the post treatment prostatectomy tissue specimens will be assessed, based upon IHC analysis following neoadjuvant PROSTVAC, ipilimumab, or the combination by flow cytometry assessment of peripheral blood mononuclear cells
Time Frame: Up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | Arm A: PROSTVAC-V/F | Arm B: Ipilimumab Monotherapy | Arm C: Combined PROSTVAC-V/F + Ipilimumab
Number analyzed (Participants) | 5 | 4 | 6
proportion of participants | 0.4 | 1.0 | 1.0

5. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: Safety analyses will be performed for all participants having received at least one dose of study drug. The investigator will use the NCI Common Terminology Criteria for Adverse Events (CTCAE) v.4.03 for reporting the number of participants with treatment-related, non-hematologic, adverse events and modified criteria for hematologic adverse events defined as having an attribute of possible, probable, or definite by toxicity and treatment group.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Arm A: PROSTVAC-V/F | Arm B: Ipilimumab Monotherapy | Arm C: Combined PROSTVAC-V/F + Ipilimumab
Number analyzed (Participants) | 5 | 4 | 6
participants
  Fatigue | 1 | 1 | 0
  Fever | 1 | 0 | 0
  Injection site reaction | 2 | 0 | 1
  Lipase increased | 1 | 0 | 0
  Pruritus | 0 | 1 | 0
  Dizziness | 0 | 0 | 1
  Skin and subcutaneous tissue disorders - Other | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Arm A: PROSTVAC-V/F | Arm B: Ipilimumab Monotherapy | Arm C: Combined PROSTVAC-V/F + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 3/4 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: PROSTVAC-V/F (N=5) | Arm B: Ipilimumab Monotherapy (N=4) | Arm C: Combined PROSTVAC-V/F + Ipilimumab (N=6)
Fatigue (General disorders) | 2 (3) | 2 (2) | 2 (2)
Injection site reaction (General disorders) | 3 (6) | 0 (0) | 3 (5)
Fever (General disorders) | 3 (3) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Lipase increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early due to low accrual, thus outcomes are not sufficiently powered for statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT02506114/Prot_SAP_000.pdf